CLINICAL TRIAL: NCT05108441
Title: Comparison of Quadriceps Femoris Measurements in Critically Ill Children, Using Bedside Ultrasound and Magnetic Resonance Imaging
Brief Title: Ultrasound and MRI Measurement of Quadriceps Femoris Muscle in Critically Ill Children
Acronym: Echo-QF-IRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1076
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Quadriceps Femoris Measurement as a Surrogate of Muscle Mass Assessment in Critically Ill Children
Keywords: Ultrasound;; Magnetic resonance imaging;; quadriceps femoris,; critically ill children
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Echo (Other): Ultrasound and magnetic resonance imaging measurements of quadriceps femoris
  Interventions: Other: Ultrasound and magnetic resonance imaging measurements of quadriceps femoris

INTERVENTIONS:
Other: Ultrasound and magnetic resonance imaging measurements of quadriceps femoris — In sedated critically ill children, quadriceps femoris thickness and cross sectional area will be measured with thigh bedside ultrasound, performed by two trained operators consecutively. These two measurements will also be made at the exact same location on a magnetic resonance imaging transverse view of the thigh, to allow comparing them to ultrasound measurements.

SUMMARY:
A vast majority of children admitted to paediatric intensive care (PICU) present with faltering growth during their admission. Muscle mass loss is an early, intense and frequent phenomenon in this setting, which is associated with impaired outcomes. Recent international guidelines recommend monitoring both nutritional status and muscle mass throughout hospital stay. Recent studies have used quadriceps femoris (QF) measurements as a surrogate for lean mass assessment, and monitored them with bedside ultrasound (QF thickness and QF cross sectional area). However, ultrasound cross sectional area inter-operator reproducibility has not been validated so far, and none of these ultrasound measurements has been validated against their gold standard i.e. magnetic resonance imaging measurements. This validation process should be conducted to allow interpreting ultrasound muscle measurements, prior to the implementation of ultrasound measurments into clinical practice.

We hypothesise that ultrasound measurements of QF thickness and cross sectional area are reliable compared to the magnetic resonance imaging gold standard, and that QF cross sectional area has a reliable inter-operator reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* critically ill children from 0 to 17 years old
* magnetic resonance imaging planned for any medical reason
* sedated child for any medical reason
* absence of parental/patient refusal to participate to the study

Exclusion Criteria:

* congenital neuromuscular disease
* no possible access to the thigh (e.g. dressing, drains, gypsum)
* anatomical anomaly of the limb, that would compromise localizing thigh landmarks (patella, groin)
* inability to obtain limb rest and/or thigh muscle decontraction
* risk induced by mobilization of the patient for ultrasound or magnetic resonance imaging purpose
* absence of social insurance

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
intraclass correlation coefficient between ultrasound measurements and magnetic resonance imaging measurements | All ultrasound measurements will be made the same day than the magnetic resonance imaging, in a 6 hour-range prior or after the magnetic resonance imaging.
  The mean of 4 measurements of quadriceps femoris thickness and the mean of 3 measurements of quadriceps femoris cross sectional area, performed by ultrasound, will be compared with the measurements means performed by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: VALLA Frédéric, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Paediatric intensive care - Hospices Civils de Lyon, Bron, Bron, France

IPD SHARING:
Plan to Share IPD: No